CLINICAL TRIAL: NCT05122260
Title: A Phase 1a Safety, Acceptability and Pharmacokinetics Study of Q-Griffithsin Intranasal Spray for Broad-spectrum Coronavirus Pre-exposure Prophylaxis: A Study of the PREVENT-COVID-19Program
Brief Title: PREVENT-COVID-19: A Q-Griffithsin Intranasal Spray
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kenneth Palmer (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kenneth Palmer, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21.0704; MCDC2006-010 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-11-01; First posted 2021-11-16 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Prevention
Keywords: COVID-19; Q-Griffithsin; Nasal Spray; Prophylactic; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — q-griffithsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Pharmacy will perform randomization and maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Q-Griffithsin (Experimental)
  Interventions: Drug: Q-Griffithsin

INTERVENTIONS:
Drug: Q-Griffithsin — intranasal spray administered as a single dose
  Arms: Q-Griffithsin
Other: Placebo — intranasal spray administered as a single dose
  Arms: Placebo

SUMMARY:
This is the first-in-human clinical study to see if a single dose of an investigational nasal spray made from a modified plant protein called Q-Griffithsin is safe, tolerated and acceptable for use by healthy adults 18 to 60 years of age.

DETAILED DESCRIPTION:
Q-Griffithsin (Q-GRFT) nasal spray is an investigational product that has broad spectrum antiviral activity. Q-GRFT is derived from Griffithsin (GRFT) a naturally occurring protein originally isolated from the red alga Griffithsia found in the South Pacific Ocean. For the purposes of this study GRFT has been genetically modified to produce a more stable compound less prone to oxidation, Q-GRFT. Q-GRFT is under study for potential therapeutic applications against several viral pathogens including HIV, herpes simplex virus type-2, and hepatitis C Q-GRFT suppresses replication of many different coronaviruses, including coronaviruses that cause the common cold, as well as Middle East Respiratory Syndrome Coronavirus (MERS-CoV) and Severe Acute Respiratory Syndrome Coronavirus type-1 (SARS-CoV) as well as Severe Acute Respiratory Syndrome Coronavirus type-2 (SARS-CoV-2).

The investigational product is a nasal spray containing Q-GRFT, and other excipients designed to optimize delivery of Q-GRFT to the nasal and naso-pharyngeal mucosa, where SARS-CoV-2 often first initiates infection.

Up to 18 healthy individuals between the ages of 18 and 60 years will be enrolled at the University of Louisville. Participants will be assigned 2:1 In a randomized and blinded fashion to receive either the Q-GRFT nasal spray or a placebo nasal spray. Participants in this study will have screening procedures including lab tests and health questions. If they are eligible for the study, they will have blood drawn for additional lab tests, have an examination of their nasal cavity by a doctor using a scope, and have nasal and throat mucus samples collected. There will be one dose of a nasal spray after the participant is randomized to their respective group. Samples will be collected at 1, 6, and 24 hours as well as 3 days after the nasal spray dose. The participant will answer questions about their quality of life, medical history and current medical status, and their experience with the study treatment. Their COVID-19 antibodies will also be checked, and they will be informed of the results. This is a phase 1 trial. The first human tests of investigational drugs or therapies occur in Phase 1 trials. Phase 1 trials are designed to determine the best dose of the study drug and to check for any potential side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 60 years at screening.
2. COVID-19 negative using Rapid antigen test at screening
3. Able and willing to provide written informed consent to take part in the study.
4. Able and willing to provide adequate information for locator purposes.
5. Availability to return for all study visits, barring unforeseen circumstances.
6. Agree not to participate in other research studies involving drugs and/or medical devices during the study period.
7. Female participants must meet the following criteria:

   * Postmenopausal or using (or willing to use) an acceptable form of contraception (e.g., barrier method, IUD, hormonal contraception, sexual abstinence, surgical sterilization, or vasectomization of male partner). If the female participant has female partners only, the method of contraception will be noted as a barrier method in the study documentation.
   * Not be pregnant at the baseline or enrollment visit
   * Not be breastfeeding at screening or intend to breastfeed during study participation per participant report
8. Willingness and ability to safely defer vaccinations until after study participation is completed.
9. Must be in general good health in the opinion of the investigator.

Exclusion Criteria:

1. Participants with ongoing moderate to severe allergic rhinitis, asthma, or history of chronic obstructive pulmonary disease (COPD) and currently suffering from chronic rhinitis or acute/chronic sinusitis.
2. Participants who report any of the following at Screening:

   1. Ongoing common cold or flu-like symptoms for 48 hours prior to the screening, including sore throat, blocked nose, runny nose, cough, and sneezing.
   2. Participants who experience moderate or severe or higher seasonal allergies, such as hay fever, (symptoms in excess of mild, intermittent nasal rhinorrhea, sneezing, or itchy/watery eyes).
   3. Non-therapeutic injection drug use in the 6 months prior to screening and recreational snorting drug use or on prescription medication/ concomitant therapy other than for contraception and antibiotics. Concomitant prescription medications may include systemic steroids, intranasal medicines, among others.
   4. Participants who are current smokers.
   5. Known Allergy to methylparaben, or propylparaben, or any ingredients of the formulated drug product.
   6. Use of systemic immunomodulatory medications (Thalidomide, Lenalidomide, Pomalidomide, Imiquimod, etc.), anticoagulants, and other drugs assessed by the site Investigator within the 4 weeks prior to the Enrollment.
   7. History of alcohol/ substance abuse within 6 months of study enrollment.
   8. History of any vaccination within the 2 weeks prior to enrollment.
   9. Participating in another research study involving drugs or medical devices within the 4 weeks prior to enrollment
   10. Having plans to relocate away from the study site area during the period of study participation
3. Has any of the following laboratory abnormalities at Screening:

   1. White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3
   2. Hemoglobin <12 g/dL for men and <11 g/dL for women.
   3. Calculated creatinine clearance >1.1 x upper limit of normal (ULN)
   4. Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 1.1 × the site laboratory ULN
   5. Total bilirubin > 1.1 x ULN
   6. ≥ +1 glucose or +2 protein on urinalysis (UA)
4. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study, or unable to comply with the study requirements. Such conditions may include but are not limited to, a current or recent history (within last 6 months) of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral disease, severe nasal septum deviation, or other condition that may cause nasal obstruction like nasal polyps or nasal/ sinus surgery in the past.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
The safety of a single exposure of Q-GRFT study product (SP) will be evaluated when administered via a nasal spray system. | 3 Weeks
  Incidence of AEs Grade 3 or higher as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events V2.1 (July 2017) will be used to determine whether the product is safe. Any emergent AEs will be discussed with the Safety Committee.
  All serious adverse events will be reported by the site investigator(s) to the Medical Monitor and IND Sponsor/Protocol Chair within 24 hours of the site becoming aware of the event.
The product acceptability will be assessed to determine its use by the participants | 3 Weeks
  The acceptability questionnaire will be filled out by the participants and provide participants' opinions on the spray characteristics, administration process, the applicator/spray design, and the use regimen, as well as the degree to which participants believe these characteristics and side-effects could pose barriers in future sustained use. The proportion of participants who report product characteristics to be considered a barrier in use, operationalized as having a rating of lower than 3 on a 5-point Likert scale, in disliking or likelihood of future barrier in use will be calculated and examined.
Pharmacokinetics of the product | 3 Weeks
  Q-GRFT Study Product (SP) concentration will be assessed in plasma, nasal, nasopharyngeal, and oropharyngeal fluids.

SECONDARY OUTCOMES:
Smell assessment will be performed to evaluate the impact of Q-GRFT SP intranasal treatment on the sensation using the University of Pennsylvania Brief Smell Identification Test (BSIT), a validated assessment of olfactory function [1]. | 3 Weeks
  The BSIT assesses an individual's ability to detect odors at a suprathreshold level. The test consists of 12 items provided in a 12-page booklet. On each page, there is a "scratch and sniff" strip embedded with a microencapsulated odorant along with 4 choice options. The scents are released by scratching the surface with a pencil, after which the participant smells the strip and chooses the odor from the four choices listed [2]. Scores range from 0-12. The BSIT has demonstrated good reliability (r=.71) and takes less than 5 minutes to complete.
  1. Doty, R.L., A. Marcus, and W. William Lee, Development of the 12-item cross-cultural smell identification test (CC-SIT). The Laryngoscope, 1996. 106(3): p. 353-356.
  2. Doty, R.L., Office procedures for quantitative assessment of olfactory function. Am J Rhinol, 2007. 21(4): p. 460-73.
Subject quality of Life (12-Item Short Form Survey (SF-12)) | 3 Weeks
  will be evaluated with the SF-12 battery of questions. Scores range from 0-100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doty RL, Marcus A, Lee WW. Development of the 12-item Cross-Cultural Smell Identification Test (CC-SIT). Laryngoscope. 1996 Mar;106(3 Pt 1):353-6. doi: 10.1097/00005537-199603000-00021. PMID 8614203
- [Background] Chen H, Cisternas MG, Katz PP, Omachi TA, Trupin L, Yelin EH, Balmes JR, Blanc PD. Evaluating quality of life in patients with asthma and rhinitis: English adaptation of the rhinasthma questionnaire. Ann Allergy Asthma Immunol. 2011 Feb;106(2):110-118.e1. doi: 10.1016/j.anai.2010.10.027. Epub 2011 Jan 8. PMID 21277512
- [Background] Doty RL. Office procedures for quantitative assessment of olfactory function. Am J Rhinol. 2007 Jul-Aug;21(4):460-73. doi: 10.2500/ajr.2007.21.3043. PMID 17882917
- [Derived] Cash E, Deitz K, Potts KL, Nabeta HW, Zahin M, Rai SN, Dryden GW, Palmer KE. Development and validation of a product acceptability questionnaire for intranasal Q-Griffithsin COVID-19 prophylaxis (SPRAY PAL). BMJ Open. 2023 Sep 12;13(9):e073735. doi: 10.1136/bmjopen-2023-073735. PMID 37699630